CLINICAL TRIAL: NCT01342471
Title: TV Commercial Stepping: Can America's Top Sedentary Activity be Made More Active
Brief Title: Physical Activity and Leisure-time Study (PALS)
Acronym: PALS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTennessee
Record Dates: First submitted 2011-04-21; First posted 2011-04-27 (Estimated); Results first posted 2012-11-09 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-10

CONDITIONS: Physical Activity; Weight
Keywords: Physical activity intervention; walking; TV; sedentary
MeSH Terms: conditions — Motor Activity; Body Weight; Sedentary Behavior | interventions — Walking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 30-min walk (Active Comparator): Instructed to use "brisk" walking (at least 30 min/day in bouts of at least 10 min) at least 5 days/week. Participants were permitted to exercise in one long bout (30 min) or divide the exercise into multiple bouts as long as the bout length was 10 min or greater.
  Interventions: Behavioral: 30-min walk
- TV commercial stepping (Experimental): Instructed to stand and "briskly" step in place, or "briskly" walk continuously around the room/house for the duration of each commercial break during at least 90 min of TV programming on at least 5 days/week. Rather than exercising continuously for at least 10-minute bouts, participants performed multiple (~9 or 10), short (~3-5 min) bouts, conveniently incorporated into their daily TV viewing time.
  Interventions: Behavioral: TV commercial stepping

INTERVENTIONS:
Behavioral: TV commercial stepping — Participants were instructed to stand and "briskly" step in place, or "briskly" walk continuously around the room/house for the duration of each commercial break during at least 90 min of TV programming on at least 5 days/week. Both conditions will receive an ankle mounted Omron pedometer, so they were able to track their steps each day. Participants were not given instructions concerning diet modification or modifying TV viewing time during a 6 month behavioral physical activity intervention
  Other Names: novel exercise prescription
  Arms: TV commercial stepping
Behavioral: 30-min walk — Participants were instructed to use "brisk" walking (at least 30 min/day in bouts of at least 10 min) at least 5 days/week. Both conditions will receive an ankle mounted Omron pedometer, so they were able to track their steps each day. Participants were not given instructions concerning diet modification or modifying TV viewing time during a 6 month behavioral physical activity intervention
  Other Names: standard physical activity prescription
  Arms: 30-min walk

SUMMARY:
Physical inactivity is a major public health problem and a primary contributing factor to the obesity epidemic. While most Americans do not meet the physical activity (PA) guidelines (30 min/day, 5 day/wk), they do report watching several hours of TV each day, and frequently site "lack of time" as a barrier for engaging in PA. The Physical Activity and Leisure-time Study examines an approach convert sedentary TV watching into active TV watching time by having adults step in place during commercials (TV commercial stepping).

DETAILED DESCRIPTION:
This randomized controlled trial will examine the effects of a PA prescription of TV commercial stepping for at least 90 min/day of TV programming, with that of walking at least 30 min/day (30 min walk) on daily step counts, TV viewing, and diet during a 24 week PA intervention. Sedentary, overweight or obese, adults will be randomly assigned to either the TV commercial stepping, or 30 min walk group during a 24-week behavioral PA intervention. Both groups will attend 8 sessions, but receive different PA goals. PA, TV watching time, diet, and anthropometric data will be collected at 0, 12, and 24 weeks. It is hypothesized that the TV commercial stepping condition will, show an equal increase in PA at 12 and 24 weeks as compared to the 30-min walk condition. Neither group is hypothesized to demonstrate changes in TV viewing time, dietary intake, or weight.

ELIGIBILITY:
Inclusion Criteria:

* 25 to 65 years of age
* BMI between 25 and 45 kg/m2
* watch ≥14 hours per week of TV
* ability to follow instructions and record data
* ability to walk 1/4 mile without stopping

Exclusion Criteria:

* history of myocardial infraction, angina, stroke, heart failure, or uncontrolled cardiac arrhythmias
* a resting blood pressure greater than 180 mm Hg systolic and/or 100 mm Hg diastolic
* other physical or medical limitations for engaging in physical activity
* no television in the home
* baseline physical activity level exceeding 7,499 steps per day as determined by the Omron pedometer
* currently participating in a program to increase PA
* intended to move outside the East Tennessee area within the time frame of the intervention
* were pregnant, lactating, less than 6 months post-partum, or planned to become pregnant during the time frame of the intervention
* unwilling to attend group intervention meetings, assessments or to complete an activity diary for the duration of the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy A Steeves, MS, Principal Investigator — University of Tennessee; Dixie Lee Thompson, Phd, Study Chair — University of Tennessee
Locations (1):
- HPER Building, 1914 Andy Holt Ave., Knoxville, Tennessee, United States

REFERENCES:
- [Derived] Steeves JA, Bassett DR, Fitzhugh EC, Raynor H, Cho C, Thompson DL. Physical Activity With and Without TV Viewing: Effects on Enjoyment of Physical Activity and TV, Exercise Self-Efficacy, and Barriers to Being Active in Overweight Adults. J Phys Act Health. 2016 Apr;13(4):385-91. doi: 10.1123/jpah.2015-0108. Epub 2015 Sep 17. PMID 26383783
- [Derived] Steeves JA, Bassett DR, Fitzhugh EC, Raynor HA, Thompson DL. Can sedentary behavior be made more active? A randomized pilot study of TV commercial stepping versus walking. Int J Behav Nutr Phys Act. 2012 Aug 6;9:95. doi: 10.1186/1479-5868-9-95. PMID 22866941

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruited by flyers and newspaper advertisements, were enrolled in a university-based PA program during the months of September through November, 2010.
Groups:
- 30-min Walk: Instructed to use "brisk" walking (at least 30 min/day in bouts of at least 10 min) at least 5 days/week. Participants were permitted to exercise in one long bout (30 min) or divide the exercise into multiple bouts as long as the bout length was 10 min or greater.
  30-min walk : Participants were instructed to use "brisk" walking (at least 30 min/day in bouts of at least 10 min) at least 5 days/week. Both conditions will receive an ankle mounted Omron pedometer, so they were able to track their steps each day. Participants were not given instructions concerning diet modification or modifying TV viewing time during a 6 month behavioral physical activity intervention
- TV Commercial Stepping: Instructed to stand and "briskly" step in place, or "briskly" walk continuously around the room/house for the duration of each commercial break during at least 90 min of TV programming on at least 5 days/week. Rather than exercising continuously for at least 10-minute bouts, participants performed multiple (~9 or 10), short (~3-5 min) bouts, conveniently incorporated into their daily TV viewing time.
  TV commercial stepping : Participants were instructed to stand and "briskly" step in place, or "briskly" walk continuously around the room/house for the duration of each commercial break during at least 90 min of TV programming on at least 5 days/week. Both conditions will receive an ankle mounted Omron pedometer, so they were able to track their steps each day. Participants were not given instructions concerning diet modification or modifying TV viewing time during a 6 month behavioral physical activity intervention
Period: Overall Study
Arm/Group | 30-min Walk | TV Commercial Stepping
Started | 29 | 29
Completed | 24 | 23
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 30-min Walk | TV Commercial Stepping | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 50.2 (9.8) | 53.8 (6.8) | 52.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity (Steps/Day)
Description: Change in pedometer measured steps per day between 0 and 6 months
Time Frame: 0 and 6 months
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | 30-min Walk | TV Commercial Stepping
Number analyzed (Participants) | 29 | 29
steps/day | 2956 (604) | 2994 (918)

2. Secondary Outcome: Total Energy Intake
Description: Change in total energy intake(kcals/day) between 0 and 6 months
Time Frame: 0 and 6 months
Measure: Mean (Standard Deviation); unit: kcals/day
Arm/Group | 30-min Walk | TV Commercial Stepping
Number analyzed (Participants) | 29 | 29
kcals/day | -354.2 (63.5) | -347.9 (256)

3. Secondary Outcome: TV Related Energy Intake
Description: Change in energy intake (kcals/day) while watching TV between 0 and 6 months
Time Frame: 0 and 6 months
Measure: Mean (Standard Deviation); unit: kcals/day
Arm/Group | 30-min Walk | TV Commercial Stepping
Number analyzed (Participants) | 29 | 29
kcals/day | -516.6 (176.4) | -282.6 (69.7)

4. Secondary Outcome: Weight
Description: Change in weight in kgs between 0 and 6 months
Time Frame: 0 and 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 30-min Walk | TV Commercial Stepping
Number analyzed (Participants) | 29 | 29
kg | -0.4 (0) | -0.7 (0.2)

5. Secondary Outcome: TV Viewing Time
Description: Change in self-reported TV viewing time per day between 0 and 6 months
Time Frame: 0 and 6 months
Measure: Mean (Standard Deviation); unit: hr/day
Arm/Group | 30-min Walk | TV Commercial Stepping
Number analyzed (Participants) | 29 | 29
hr/day | -1.4 (0.6) | -1.2 (0)

ADVERSE EVENTS:
Arm/Group | 30-min Walk | TV Commercial Stepping
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

LIMITATIONS AND CAVEATS:
Small sample size, disproportionate female gender participation, and limited ethnic diversity. No follow up after 6 months. No control group, that received no intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes